CLINICAL TRIAL: NCT00309907
Title: Soluble Tumor Necrosis Factor Receptor: Enbrel® (Etanercept) for the Treatment of Acute Non-Infectious Pulmonary Dysfunction (Idiopathic Pneumonia Syndrome) Following Allogeneic Stem Cell Transplantation
Brief Title: Etanercept in Treating Young Patients With Idiopathic Pneumonia Syndrome After Undergoing a Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASCT0521; NCI-2009-00429 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-PBMTC-SUP051 (Other: Children's Oncology Group); COG-ASCT0521 (Other: Children's Oncology Group); CDR0000456407 (Other: Clinical Trials.gov); U10CA098543 (NIH)
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Results first posted 2014-02-14 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-02

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Blastic Phase Chronic Myelogenous Leukemia; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Chronic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Disseminated Neuroblastoma; Juvenile Myelomonocytic Leukemia; Previously Treated Childhood Rhabdomyosarcoma; Previously Treated Myelodysplastic Syndromes; Pulmonary Complications; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Neuroblastoma; Recurrent Wilms Tumor and Other Childhood Kidney Tumors; Recurrent/Refractory Childhood Hodgkin Lymphoma; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Neuroblastoma; Wilms Tumor; Recurrence | interventions — Etanercept; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etanercept and corticosteroid therapy (Experimental): Patients receive etanercept IV (dose 0.4 mg/kg- max 25 mg) over 30 minutes on day 0 and subcutaneously (dose 0.4 mg/kg- max 25 mg) on days 3, 7, 10, 14, 17, 21, and 24. Treatment continues in the absence of an infectious pathogen, disease progression, or unacceptable toxicity. Patients also receive methylprednisolone (or corticosteroid equivalent) IV (dose 2.0 mg/kg/day) on days 0-2 and then orally with a taper beginning day 7. Dose on days 7-20 (1.0 mg/kg/day), days 21-34 (0.5 mg/kg/day), days 35-48 (0.25 mg/kg/day) and days 49-56 (0.25 mg/kg/every other day) discontinuing on day 56.
  Interventions: Biological: etanercept; Drug: methylprednisolone

INTERVENTIONS:
Biological: etanercept — Given IV and subcutaneously
  Other Names: Enbrel; ETN; TNFR:Fc; Tumor Necrosis Factor Receptor IgG Chimera
Drug: methylprednisolone — Given IV and orally
  Other Names: Depo-Medrol; Medrol; MePRDL; Solu-Medrol; Wyacort

SUMMARY:
This phase II trial is studying how well etanercept works in treating young patients with idiopathic pneumonia syndrome after undergoing a donor stem cell transplant. Etanercept may be effective in treating patients with idiopathic pneumonia syndrome after undergoing a donor stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate, defined as survival and complete discontinuation of supplemental oxygen at day 28, in pediatric patients with acute noninfectious pulmonary dysfunction (idiopathic pneumonia syndrome [IPS]) after undergoing allogeneic stem cell transplantation treated with etanercept.

SECONDARY OBJECTIVES:

I. Estimate the day 56 survival rate in patients treated with this drug. II. Determine the overall survival distribution in patients treated with this drug.

III. Determine the pulmonary response, as defined as the time to discontinuation of supplemental oxygen, in patients treated with this drug.

IV. Evaluate the toxicity of etanercept therapy in patients with IPS. V. Evaluate levels of pro-inflammatory cytokines, in both bronchoalveolar lavage (BAL) fluid and serum, in patients with IPS.

VI. Describe C-reactive protein (CRP) levels at baseline, day 7, 14, 21, and 28 and their association with response in patients with IPS.

OUTLINE: This is an open-label, nonrandomized, multicenter study.

Patients receive etanercept IV over 30 minutes on day 0 and subcutaneously on days 3, 7, 10, 14, 17, 21, and 24. Treatment continues in the absence of an infectious pathogen, disease progression, or unacceptable toxicity. Patients also receive methylprednisolone (or corticosteroid equivalent) IV on days 0-2 and then orally with a taper until day 56.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute, noninfectious idiopathic pulmonary dysfunction (IPS) as defined by the following:

  * Evidence of diffuse lung injury occurring within the first several months after hematopoietic stem cell transplantation for which an infectious etiology is not identified. To meet the criteria for IPS there must be:

    * Evidence of widespread alveolar injury

      * Diffuse multi-lobar infiltrates on chest x-ray or CT scan
      * Evidence for abnormal respiratory physiology based upon 1 of the following:

        * Room air oxygen saturation < 93%
        * Supplemental oxygen required to maintain an oxygen saturation ≥ 93%
    * Absence of active lower respiratory tract infection, defined as Bronchoalveolar lavage (BAL)-negative for infection based on one of the following:

      * Gram stain, fungal stain, acid-fast bacilli stain
      * Bacterial culture (a quantitative culture ≥ 10^4 colony-forming units/mL is considered positive)
      * Fungal culture
      * Mycobacterial culture
      * Viral culture (respiratory syncytial virus [RSV], parainfluenza, adenovirus, influenza A and B, and cytomegalovirus [CMV])

        * If direct fluorescent antibody (DFA) screening is performed on BAL, it must be negative for all viruses listed above
      * Pneumocystis carinii pneumonia by polymerase chain reaction (PCR), DFA stain, or cytology
  * Evidence of bilateral pulmonary infiltrates (on chest radiograph)
  * Patients may have diffuse alveolar hemorrhage (DAH) or peri-engraftment respiratory distress syndrome (PERDS)
  * Presence of "mixed oral flora," "rare Candida species," or the presence of a Penicillium species reported on BAL fluid analysis allowed
  * A radiographic finding of pulmonary edema does not exclude the diagnosis of IPS, provided the other criteria have been met and provided the treating physician concludes by clinical (or echocardiographic) criteria that the pulmonary edema is not secondary to cardiac dysfunction or iatrogenic fluid overload
* Patients must require supplemental oxygen
* Must have undergone an allogeneic bone marrow, cord blood, or peripheral blood stem cell transplantation within the past 120 days

  * There are no restrictions based upon underlying disease, donor source, the degree of HLA match, the intensity of the pre-transplant conditioning regimen, or the use of a prior donor leukocyte infusion
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No documented invasive fungal or systemic viral infection within the past 14 days

  * Patients with asymptomatic viruria allowed
* No signs of CMV reactivation (by CMV, PCR, antigenemia, or shell vial culture) within the past 14 days
* No sepsis syndrome or hypotension that requires inotropic support (except dopamine < 5mcg/kg/minute)
* No documented bacteremia within the past 48 hours

  * Persistent fever allowed
* No evidence of cardiac failure by clinical or echocardiographic findings
* No known hypersensitivity to etanercept
* No known history of tuberculosis (Tb) or prior Tb exposure
* No prior chronic hepatitis B or hepatitis C infection
* Concurrent treatment for acute or chronic GVHD allowed
* More than 14 days since prior etanercept
* More than 7 days since prior investigational drug trials (phase I, II, or III) for the treatment of acute graft-versus-host disease (GVHD)
* Not on mechanical ventilation for > 48 continuous hours prior to study entry
* Must not be receiving > 2 mg/kg/day of methylprednisolone or corticosteroid equivalent within 24 hours of study entry
* Concurrent continuous veno-venous hemofiltration or hemodialysis allowed

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2006-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Yanik, MD, Principal Investigator — Children's Oncology Group
Locations (26):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Oncology Group, Arcadia, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Childrens Memorial Hospital, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Indiana University Medical Center, Indianapolis, Indiana
  - Children's Hospital-Main Campus, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Etanercept and Corticosteroid Therapy
Started | 39
Completed | 19
Not Completed | 20
Not completed — Death | 4
Not completed — Physician Decision | 1
Not completed — Ineligible | 11
Not completed — Major infectious event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept and Corticosteroid Therapy
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 11 [1 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 22
  More than one race | 0
  Unknown or Not Reported | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35
  Canada | 2
  Sri Lanka | 1
  Saudi Arabia | 1

OUTCOME MEASURES:

1. Primary Outcome: Response of IPS (Idiopathic Pneumonia Syndrome) to Etanercept Plus Corticosteroid Therapy by Day 28.
Description: Response to therapy is defined as survival to Day 28 of study, PLUS complete discontinuation all supplemental oxygen support by Day 28 of study. Subjects must be able to remain off all supplemental oxygen support for > 72 consecutive hours. Subjects who discontinue supplemental oxygen within the last 72 hours of the observation period will be followed until they have completed 72 consecutive hours off oxygen or failed prior to assessing response.
Time Frame: At day 28
Population: Analysis population includes all patients who are eligible and had sufficient data to evaluate response. Eleven ineligible patients are excluded.
Measure: Number; unit: participants
Arm/Group | Etanercept and Corticosteroid Therapy
Number analyzed (Participants) | 28
participants
  With Response | 20
  Without Response | 8

2. Secondary Outcome: Survival Rate
Description: Estimated Day 56 survival rate following initiation of etanercept + corticosteroid therapy for patients with IPS.
Time Frame: Up to day 56
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Etanercept and Corticosteroid Therapy: Regimen A
Arm/Group | Etanercept and Corticosteroid Therapy
Number analyzed (Participants) | 28
percentage of participants | 75 [55 to 87]

3. Secondary Outcome: Estimate Percentage Pulmonary Response in Patients With IPS Treated With Etanercept + Corticosteroid Therapy
Description: Pulmonary response is defined as alive & come off of oxygen .
Time Frame: up to day 56
Population: Total of 28 patients are evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept and Corticosteroid Therapy
Number analyzed (Participants) | 28
percentage of participants | 74

4. Secondary Outcome: Toxicity of Etanercept Plus Corticosteroid Therapy Using the Common Terminology Criteria Version 4.0
Description: Grade 3-5 organ toxicities attributable to etanercept.
Time Frame: Up to 56 days
Population: 28 patients evaluable for this outcome.
Measure: Number; unit: Patients
Arm/Group | Etanercept and Corticosteroid Therapy
Number analyzed (Participants) | 28
Patients | 0

5. Secondary Outcome: Plasma Cytokine IL6 Level
Description: Estimated mean and standard error of IL6 level
Time Frame: From baseline to days 7 and 28
Population: Plasma samples were available for biomarker analysis in 26 patients. The data were intended to be analyzed for all subjects, therefore, combined result is reported.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Etanercept and Corticosteroid Therapy
Number analyzed (Participants) | 26
pg/ml
  Baseline | 205.2 (58)
  Day 7 | 28.8 (4.4)
  Day 28 | 23.1 (3.5)

6. Secondary Outcome: C-reactive Protein Levels
Description: Estimated mean and standard deviation
Time Frame: From baseline to days 7, 14, 21, and 28
Population: The data for baseline were intended to be analyzed for all subjects, therefore, combined result is reported. The data for Days 7, 14, 21 and 28 were intended to be analyzed by subgroups of subjects as pre-specified in the study protocol, therefore combined result us not reported for Etanercept + corticosteroid therapy treatment arm.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Etanercept and Corticosteroid Therapy
Number analyzed (Participants) | 28
mg/dL
  Baseline: number analyzed (Participants) | 24
  Baseline | 28.1 (59.1)
  Day 7 Non Responders: number analyzed (Participants) | 12
  Day 7 Non Responders | 5.4 (11.4)
  Day 7 Responders: number analyzed (Participants) | 10
  Day 7 Responders | 1.8 (1.9)
  Day 14 Non Responders: number analyzed (Participants) | 10
  Day 14 Non Responders | 4.9 (11.1)
  Day 14 Responders: number analyzed (Participants) | 8
  Day 14 Responders | 1 (1.1)
  Day 21 Non Responders: number analyzed (Participants) | 7
  Day 21 Non Responders | 10.7 (14.3)
  Day 21 Responders: number analyzed (Participants) | 12
  Day 21 Responders | 1.6 (2.4)
  Day 28 Non Responders: number analyzed (Participants) | 5
  Day 28 Non Responders | 19.6 (29.7)
  Day 28 Responders: number analyzed (Participants) | 14
  Day 28 Responders | 5.3 (16.1)

ADVERSE EVENTS:
Description: Eleven ineligible patients are not reported in the adverse events.
Arm/Group | Etanercept and Corticosteroid Therapy
Serious Adverse Events (participants affected / at risk) | 5/28
Other Adverse Events (participants affected / at risk) | 6/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept and Corticosteroid Therapy (N=28)
Acute kidney injury (Renal and urinary disorders) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Alkalosis (Metabolism and nutrition disorders) | 1
Blood bilirubin increased (Investigations) | 1
Death NOS (General disorders) | 1
Esophageal hemorrhage (Gastrointestinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 1
Multi-organ failure (General disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept and Corticosteroid Therapy (N=28)
Acute kidney injury (Renal and urinary disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Creatinine increased (Investigations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
White blood cell decreased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No